CLINICAL TRIAL: NCT07195890
Title: Evaluation of the Effectiveness of Teen Mental Health First Aid in Secondary School Students in Hong Kong
Acronym: tMHFA-HK
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TN Foo Centre for Positive Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TNFoo Centre, MHAHK
Record Dates: First submitted 2025-09-14; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Healthy Subjects (HS)
Keywords: teen mental health first aid; knowledge of mental illness; attitude towards the mentally ill; help seeking behavior
MeSH Terms: conditions — Help-Seeking Behavior

STUDY DESIGN:
Intervention Model Description: A course of teen Mental Health First Aid will be provided to the study subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- teen Mental Health First Aid course (Other): A study group of participants receiving the t MHFA course and a control group without the course
  Interventions: Other: A course of teen Mental Health First Aid to be provided to participants

INTERVENTIONS:
Other: A course of teen Mental Health First Aid to be provided to participants — The teen Mental Health First Aid course consists of three sessions developed in Mental Health First Aid in Australia. It has been translated and attuned to the Chinese in Hong Kong.

SUMMARY:
Mental health problems in adolescents are on the rise worldwide especially after COVID -19 pandemic. Early detection and intervention should help to reduce the adverse impact of the mental illness on the adolescent. Yet the adolescent may not be able to recognize mental illness, have stigma against the mentally ill and mental health services, and may not seek help even with mental illness. The local situation in Hong Kong has been reviewed and presented in a separate article (Lai, 2024). The high prevalence of psychiatric conditions in Hong Kong adolescents has been reported (Chan et al, 2025). Teen Mental Health First Aid (t MHFA) is a course developed in Australia for the promotion of mental health literacy including awareness of mental illness, reduction of stigmatizing attitudes towards people with mental illness, and increase in appropriate help-seeking attitude and behavior among adolescents with emerging mental health problems (Hart, 2016). Mental Health Association of Hong Kong has run the mental health first aid courses in Hong Kong since 2004. The teen MHFA course has been translated and attuned to the local context recently. MHAHK has been funded by the Hong Kong Jockey Club in a two-year project in the development of a quality mental health campus in twenty secondary schools. In the project there will be mental health education programs for teachers, parents and students and mental health promotion activities in the schools. Teen MHFA will be provided to the students in the schools. It is a three-hour course separated into three separate sessions taught by trained instructors of MHAHK.

The study will obtain a baseline information about the awareness of mental illness, the attitude towards the mentally ill and help seeking behavior of secondary school students, and to verify the effectiveness of the teen MHFA course in promotion of mental health literacy of the participants, and to guide the further refinement and development of an effective course. It is hoped that the teen MHFA course can be available to all secondary schools and can help adolescents to develop appropriate mental health literacy at this important phase of development before reaching adulthood.

DETAILED DESCRIPTION:
The study is an initial evaluation of the t MHFA in secondary school students in Hong Kong. Teen MHFA was initially evaluated in Australia (Hart et al, 2016). The study is a replication of the initial study by Hart et al but followed a quasi-experimental design as in the study of MHFA done in MHAHK (Wong et al, 2015).

Secondary school students from Form 4 to Form 6 arranged by the individual schools to attend the teen Mental Health First Aid course in the Quality Mental Health Campus Project will be invited to participate in the study as study subjects. Similar numbers of students from the same forms and in the same schools not attending the course will be invited to be the control. Consent from parents is to be obtained. An estimate of about 250 students with consent from parents and an equal number of students as the control group are included to allow statistical analysis. A self-administered questionnaire used in the Australian study of teen Mental Health First Aid will be translated, adopted to the local context and used in the study. The questionnaire in digital form will be administered to the study subjects within three weeks before the course as a baseline survey, immediately after the course as the first post-course survey, and about three months later as the second post-course survey. For the control group survey will be administered around the same time of baseline survey for study subjects and then three months after the baseline survey. The questionnaire is expected to be completed within 15 minutes.

The data are compiled for basic information about the study subjects and control subjects, and to verify any difference between the study subjects and the control subjects. The baseline information about awareness of mental illness, the attitude towards the mentally ill and help seeking behavior of adolescents will be compiled. The null hypothesis is to be applied to the statistical analysis in verifying the changes after the intervention in the study subjects and whether the changes are sustained after an interval of three months. Content analysis of open-ended responses including satisfaction and comments about the teen MHFA course will be done by the investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Students
2. Form 4 to 6
3. Mainstream Chinese secondary schools in Hong Kong
4. Schools sponsoring teen Mental Health First Aid courses to students

Exclusion Criteria:

1. Students unable to give consent
2. Parents/guardians unable to give consent

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge of mental illness, attitude towards the mentally ill and help seeking behavior | A pre-test questionnaire is within three weeks before the course of teen MHFA. The first post-test questionnaire is immediately after the course of teen MHFA. The second post-test questionnaire is three months after the course.
  A questionnaire with two case vignettes is administered to a subject to assess the knowledge of mental illness, attitude towards the mentally ill, and the help seeking behavior.
Knowledge of mental illness, attitude towards the mentally ill and help seeking behavior | Pre-test is done within the week before the t MHFA course. 1st post test done immediately after the course. 2nd post test to be done after 3 months. Control group will have tests done around the time of pre-test and 3 months later.
  A self-administered questionnaire used in the Australian study of teen Mental Health First Aid will be translated, adopted to the local context and used in the study. The questionnaire in digital form will be administered to the study subjects within three weeks before the course as a baseline survey, immediately after the course as the first post-course survey, and about three months later as the second post-course survey. For the control group survey will be administered around the same time of baseline survey for study subjects and then three months after the baseline survey.
Knowledge of mental illness, attitude towards the mentally ill and help seeking behavior for mental illness | Pre-test is done in the week before the intervention. 1st post test is immediately done after the course.
  The participants and control subjects will be measured with a questionnaire developed in Mental Health First Aid in Australia
knowledge and attitude towards mental illness and the mentally ill, and help seeking behavior. | pre-test is done in the week before the course of teen Mental Health First Aid, and 1st post test will be done immediately after the course.
  questionnaire is developed in Australia for teen Mental Health First Aid

CONTACTS AND LOCATIONS:
Locations (1):
- TN Foo Centre for Positive Mental Health, Mental Health Association of Hong Kong, Hong Kong, Hksar, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The information of the individual participants will be kept confidential. Only the collective data will be analyzed.

REFERENCES:
- [Background] Wong, D. F. K., Lau, Y., Kwok, S., Wong, P. (2015). Evaluating the effectiveness of mental health first aid programme for Chinese people in Hong Kong. Research on Social Work Practice, 27(1). doi:10.1177/1049731515585149
- [Background] Lai, B. (2024). Promotion of Mental Health Literacy and Help-Seeking Behaviour of Adolescents with Mental Health Problems - The Local Perspective. Hong Kong Journal of Mental Health 2024, 50(2), 40-49.
- [Background] Hart LM, Mason RJ, Kelly CM, Cvetkovski S, Jorm AF. 'teen Mental Health First Aid': a description of the program and an initial evaluation. Int J Ment Health Syst. 2016 Jan 19;10:3. doi: 10.1186/s13033-016-0034-1. eCollection 2016. PMID 26788123
- [Background] Chan SSM, Wong OWH, Hussain S, Tsoi KKF, Ma KKY, Chau SWH, Ma SL, Lai KYC, Chu WCW, Lo HHL, Ho SWS, Leung CC, Yiu KKL, So SHW, Sham PC, Hung SF, Leung PWL. Twelve-month prevalence of DSM-5 mental disorders and the psychosocial correlates- a child and adolescent psychiatric epidemiologic survey in Hong Kong SAR. Lancet Reg Health West Pac. 2025 Mar 29;57:101533. doi: 10.1016/j.lanwpc.2025.101533. eCollection 2025 Apr. PMID 40236269

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT07195890/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT07195890/ICF_001.pdf